CLINICAL TRIAL: NCT03668587
Title: Feasibility and Security of a Rapid Rule-out and rule-in Troponin Protocol in the Management of NSTEMI in an Emergency Departement.
Acronym: ICTUS
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC18_0215
Record Dates: First submitted 2018-08-21; First posted 2018-09-12 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Troponin Protocol — Feasibility and security of a rapid rule-out and rule-in troponin protocol in the management of NSTEMI in an Emergency Departement.

SUMMARY:
Management of NSTEMI in emergency departements represent 10% of the global activity. Since the the last European Society of Cardiology recommendation the use of an 1 hour rule-in and rule-out protocol is recommended combined with high-sensitivity troponin. But studies show 3% of the patients are false negative using this protocol. This study aims at analysing the feasibility of this protocol in an Emergency Departement and the security of this protocol if combined with a pre-troponin probability score.

DETAILED DESCRIPTION:
Chest pain is a frequent reason for consultation in emergency departments. Among cardiological causes, quickly diagnosing NSTEMI optimize patient treatment. To do this, the European Society of Cardiology, proposed in 2015 an one hour rule-in rule out troponin dosage based protocol. These recommendations should allow a faster diagnosis of NSTEMI but also a rule-out of patients with a low to moderate clinical probability of coronary heart disease. It could also improve efficiency in emergency departements decreasing the length of stay for patient consulting for acute chest pain allowing use of medical and para medical time for other patients. But the studies on which thoserecommendations are based show up to 3% of false negative, which could lead to a higher mortality rate for those patients even if this issue hasn't been address yet. Furthermore, the tight schedule in which a blood sample need to be withdraw, analyzed and taken knowledge of by the doctor could be an obstacle to the feasibility of such protocol in emergency departments usually overwhelmed with patients. The aim of this monocentric prospective study is to assess how a pre-troponin clinical probability of NSTEMI allowing risk stratification could decrease the false negative rate of this protocol insuring safetiness in its use. The secondary objective is to assess the feasibility of such protocol in an emergency department with high patient flow.

ELIGIBILITY:
Inclusion Criteria:

* Patient with troponin dosage in a suspected NSTEMI.

Exclusion Criteria:

* Under 18 years old
* Respiratory rate over 30 per min
* SpO2 under 92%
* Tachycardia over 110 per min
* Bradycardia under 40 per min
* Fever over 38°5C,
* Anemia under 10 g/dL
* Acute intoxication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with troponin dosage in a suspected NSTEMI.
Sampling Method: Probability Sample
Enrollment: 1099 (Actual)
Dates: Start 2018-09-29 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Mortality at 30 day succeeding discharge | 30 days
  After hospital discharge, patients are contacted after 30 day by telephone calls or in written form. Information regarding death are furthermore obtained from the national registry on mortality, the hospital's diagnosis registry, and the family physician's records.

SECONDARY OUTCOMES:
Respect of the 1-hour rule-in and rule-out protocol | 24 hours
  Respect of the 1-hour protocol is assessed by the the respect of the dosage's time frame.
Respect of the 1-hour rule-in and rule-out protocol | 24 hours
  Respect of the 1-hour protocol is assessed by the number of troponin dosage
Respect of the 1-hour rule-in and rule-out protocol | 24 hours
  Respect of the 1-hour protocol is assessed by the patient's discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France